CLINICAL TRIAL: NCT03496896
Title: Transition cAre inteRvention tarGeted to High-risk patiEnts To Reduce rEADmission (TARGET-READ)
Brief Title: Transition cAre inteRvention tarGeted to High-risk patiEnts To Reduce rEADmission
Acronym: TARGET-READ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); University of Bern (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018-00084
Record Dates: First submitted 2018-04-04; First posted 2018-04-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Patient Readmission
Keywords: Randomized Controlled Trial; Patient readmission; Patient transfer; Health care utilization; Prognosis; Multimorbidity; Internal medicine
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the intervention, it will be not possible to blind patients and nurses providing the TARGET intervention. However, treatment allocation in the database will be coded and the study nurses collecting the outcomes or working on data cleaning and the statistician performing the analysis will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "TARGET" intervention (Experimental): The intervention group will receive a standardized transition care intervention by a trained nurse composed of a pre-discharge component and 2 post-discharge follow-up phone calls 3 days and 14 days after discharge.
  Interventions: Other: TARGET
- Control (No Intervention): The group control will receive usual care without additional intervention.

INTERVENTIONS:
Other: TARGET — The pre-discharge component includes mainly patient information, medication reconciliation, patient education, planning of a first post-discharge primary care physician visit with a timely discharge summary sent to the primary care physician. Two follow-up phone calls are made by a nurse, at D3 and D14, and include the assessment of the general health condition, the verification of the follow-up care plan, a reinforcement of the patient education, and review with the patient of the medication list with assessment of potential adverse drug events.
  Arms: "TARGET" intervention

SUMMARY:
Hospital rehospitalizations within 30 days are frequent and represent a burden for the patients, but also for the entire health care system. This study evaluates the impact of an intervention targeted to high-risk medical patients in order to reduce their risk of rehospitalization. Half of the patients will receive a set of interventions before and after their hospital discharge, while the other half will receive usual care.

DETAILED DESCRIPTION:
Background: Hospital readmissions within 30 days are frequent, with rates varying usually between 12 and 20%. Is it therefore recognized as important to improve the quality of the transition of care period in order to avoid as much as possible hospital readmissions. There are however still several gaps in current knowledges. First, most trials to reduce hospital readmission have been performed on specific patient populations such as patients with diabetes or heart failure, and therefore the findings may not be well generalizable to other high-risk population. Second, while some specific interventions have been showed to reduce readmission, these were complex and resources demanding, and no trial targeted these interventions to the patients who are most likely to benefit for better effectiveness, using a widely validated prediction tool, such as the "HOSPITAL" score. Finally, most studies tested unimodal interventions instead of more promising multimodal interventions.

Specific aim: the goal of this proposal is to evaluate the effect of a multimodal transitional care intervention prioritized to higher-risk medical patients on the composite of 30-day unplanned readmissions and death.

Methods: the investigators will conduct a multicenter randomized controlled trial in medical inpatients discharged home or nursing home, who are identified as having a higher risk for 30-day readmission. Risk of readmission will be predicted using the simplified HOSPITAL score, which includes 6 variables routinely available before hospital discharge and which has been previously validated in more than 200,000 patients across 6 countries in its original version, and in nearly 120,000 patients in its simplified version. Patients will be randomly assigned to the intervention group or usual care group. The primary outcome will be the first 30-day unplanned readmission or all-cause mortality. The primary analysis will be a comparison between two groups according to the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients planned to be discharged home/nursing home from a medical department.
* Hospital stay of at least 24 hours.
* Patient at higher risk of 30-day readmission based on the simplified HOSPITAL score.

Exclusion Criteria:

* Previous enrolment in this trial.
* Patient is not living in the country in the next 30 days.
* No phone to be reached at.
* Not speaking the local language.
* Refusal to participate, or unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1393 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
30-day unplanned readmission or death | 30 days after hospital discharge
  Number of patients who have a first unplanned readmission or die within 30 days after discharge (Composite endpoint).

SECONDARY OUTCOMES:
First 30-day unplanned readmission | 30 days after hospital discharge
  Number of patients who have a first unplanned readmission (individual components of the primary composite outcome)
30-day mortality | 30 days after hospital discharge
  Number of patients who die (individual components of the primary composite outcome).
Time to first unplanned readmission or death | Within 30 days after hospital discharge
  Number of days between hospital discharge and first unplanned readmission or death.
Patient's perspective (satisfaction) on quality of transition of care between hospital and home | 30 days after hospital discharge
  Proportion of patients who are responding positively to all 3 items of the Three-Item Care Transition Measure (CTM-3)
Post-discharge health care utilization 1 | 30 days after hospital discharge
  Total number of readmission(s)
Post-discharge health care utilization 2 | 30 days after hospital discharge
  Total number of days of hospitalizations within 30 days
Post-discharge health care utilization 3 | 30 days after hospital discharge
  Number of emergency room visits
Post-discharge health care utilization 4 | 30 days after hospital discharge
  Number of primary care provider visits
Main cause of readmission or death | 30 days after hospital discharge
  Proportion of most frequent main diagnosis for the readmission
Costs of readmission | 30 days after hospital discharge
  Total costs of the rehospitalization in Swiss Francs (CHF)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Donzé, MD, MSc, Principal Investigator — Bern University Hospital
Locations (4):
- Switzerland (4):
  - Centre hospitalier Bienne, Biel/Bienne, Canton of Bern
  - Hôpital cantonal Fribourg, Fribourg
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne
  - Hôpital neuchâtelois, Neuchâtel

REFERENCES:
- [Derived] Donze J, John G, Genne D, Mancinetti M, Gouveia A, Mean M, Butikofer L, Aujesky D, Schnipper J. Effects of a Multimodal Transitional Care Intervention in Patients at High Risk of Readmission: The TARGET-READ Randomized Clinical Trial. JAMA Intern Med. 2023 Jul 1;183(7):658-668. doi: 10.1001/jamainternmed.2023.0791. PMID 37126338

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT03496896/SAP_000.pdf